CLINICAL TRIAL: NCT03060278
Title: Smartphone-delivered Automated Video-assisted Smoking Treatment for Patrons of a Food Resource Center: Project AVAST - FRC
Brief Title: Smartphone-delivered Automated Video-assisted Smoking Treatment for Patrons of a Food Resource Center
Acronym: AVAST-FRC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7277
Record Dates: First submitted 2017-01-10; First posted 2017-02-23 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Smoking Cessation
Keywords: smoking cessation, food pantry
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Participants randomized to Standard Treatment will receive a smartphone with active service, brief advice to quit smoking (self-help materials), an 8-week supply of nicotine replacement therapy (patches), and provided 5 proactive phone counseling sessions by a trained Certified Tobacco Treatment Specialist.
  Interventions: Behavioral: Self-help materials; Drug: nicotine patch; Behavioral: Counseling
- Automated Treatment (Experimental): Participants randomized to Automated Treatment will receive smartphone-delivered automated treatment that will provide tailored smoking cessation treatment by way of video clips, text and graphical messages. Participants will receive notifications on study provided smartphone once a week for an 8-week treatment period. Content delivered will be specific to the participants smoking status and motivation to quit.
  Interventions: Behavioral: Self-help materials; Drug: nicotine patch; Other: Smartphone-delivered automated treatment

INTERVENTIONS:
Behavioral: Self-help materials — Self-help smoking cessation materials.
Drug: nicotine patch — Participants who smoke >10 cigarettes per day will receive 4 weeks of 21 mg, 2 weeks of 14 mg and 2 weeks of 7 mg nicotine patches. Participants who smoke < 10 cigarettes per day will receive 6 weeks of 14 mg and 2 weeks of 7 mg nicotine patches.
Other: Smartphone-delivered automated treatment — Tailored video clips, text and graphical messages delivered automatically each week to the participant.
  Arms: Automated Treatment
Behavioral: Counseling — Proactive phone counseling with a Certified Tobacco Treatment Counselor
  Arms: Standard Treatment

SUMMARY:
The proposed pilot study seeks to address the smoking cessation treatment needs of underserved smokers with limited resources by evaluating the feasibility and preliminary efficacy of a smartphone delivered automated video-assisted smoking treatment (AVAST). AVAST will enable smoking cessation treatment content to be presented with voice/audio, images, videos, and text in an interactive, structured format anytime and anywhere. Participants will be recruited from the Urban Mission, a non-profit food and resource center that serves approximately 20,000 people each year in the Oklahoma City metro area.

DETAILED DESCRIPTION:
Smoking remains the leading cause of preventable morbidity and mortality in the United States,1-3 with tobacco use accounting for more deaths each year than the combined deaths attributable to alcohol, other drugs, homicide, suicide, motor vehicle accidents, and sexual behavior.4 While smoking cessation decreases the risk of lung cancer, other cancers, heart attack, stroke, and chronic lung disease,5 smoking quit rates are low. Approximately 40-50% of adult daily smokers make a quit attempt each year, but less than 14% of those smokers are able to maintain abstinence for even a single month.6 Individuals with low socioeconomic status are far more likely to smoke and are less successful at quitting.7-9 Thus, smoking is a critically significant behavioral risk factor that contributes to social disparities in the incidence and mortality of disease.10-15 Data indicate that smokers with higher socioeconomic status are more likely than those with lower socioeconomic status to use effective resources for quitting smoking, which appears to partially explain their higher cessation rates.16 Therefore, efficiently connecting underserved smokers with limited resources to efficacious tobacco cessation programs that are easily accessible is crucial for disease prevention and the elimination of health disparities.

Food security is defined by the United States Department of Agriculture (USDA) as having consistent, dependable access to enough food for all household members to lead an active, healthy life.17 In 2014, 14% of US households were classified as food insecure,17 a condition that describes limited or uncertain access to nutritionally adequate, personally acceptable, and safe foods.18 National studies indicate food insecurity within low-income households is associated with hypertension (24.6%), self-reported hyperlipidemia (43.3%), diabetes (10.2%), and smoking (35%).19 Emerging data suggests populations accessing foods at food pantries fare worse compared to the general low income, food insecure population, with self-reported hypertension (65.4%) and diabetes (25.9%) being notably higher.20

Participants (n=20) will be randomized to one of two treatment conditions: 1) Standard Treatment (ST; n=10) or Automated Treatment (AT; n=10). In the ST condition, research staff will provide participants with in- person brief advice to quit and enroll them in a proactive telephone counseling program for smoking cessation. This ST approach mirrors the Ask Advise Connect (AAC) approach that our team has previously developed and implemented in numerous clinic settings.21,22 ST will be evaluated against AT, the fully automated AVAST approach. In the AT condition, smokers will be provided with brief in-person advice to quit and be enrolled in a fully automated and interactive smartphone-based treatment program that comprises interactive text messaging, images and audio/video clips. Participants in both treatment conditions will be provided with nicotine replacement therapy (NRT) in the form of transdermal patches. The goal of this pilot project is to establish the preliminary efficacy and feasibility of AT. Data collected in the pilot will then be used to support the submission of a NIH R01 application (or equivalent), and to determine if AT performs no worse than the more resource intensive ST approach. If lack of inferiority is established in the larger project, the AT approach will be readily scalable; easily implemented by community-based clinics and organizations; and offer an efficient way to allocate limited public health resources to tobacco control interventions.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years
* Smoked >/= 100 cigarettes in a lifetime
* English speaking
* Currently smoking 5 or more cigarettes per day
* Willing to make a quit attempt within 1 week of enrollment
* Patron of the Urban Mission Food Resource Center

Exclusion Criteria:

* History of medical condition that precludes the use of nicotine replacement therapy
* Current use of smoking cessation medications
* Pregnant or nursing
* Enrolled in another smoking cessation study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Smoking Status | 3-Month Follow-Up
  Biochemically verifying smoking status on all participants by collecting an expired carbon monoxide breath sample.

SECONDARY OUTCOMES:
Participant satisfaction with treatment | 3-Month Follow-Up
  The investigators will use the Client Satisfaction Questionnaire to evaluate participant satisfaction.
Dropout rate | 3-Month Follow-Up
  The investigators will assess the number of participants who dropped out of the study.
Intervention delivery rate | 3-Month Follow-Up
  The investigators will assess the number of sessions completed by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, DrPH, Principal Investigator — OUHSC
Locations (1):
- Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No